CLINICAL TRIAL: NCT04221399
Title: A Single- and Multiple-Dose Clinical Study to Evaluate Pharmacokinetics and Pharmacodynamics of DWP16001 Following Oral Dose in Type 2 Diabetes Patients With Renal Impairment
Brief Title: Type 2 Diabetes Patients With Renal Impairment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001103
Record Dates: First submitted 2019-12-17; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP16001 Single dose (Experimental): Single dose
  Interventions: Drug: DWP16001
- DWP16001 Multiple dose (Experimental): Up to 7 days
  Interventions: Drug: DWP16001

INTERVENTIONS:
Drug: DWP16001 — Tablets, Oral, Once daily, Single dose
  Arms: DWP16001 Single dose
Drug: DWP16001 — Tablets, Oral, Once daily, Multiple dose
  Arms: DWP16001 Multiple dose

SUMMARY:
The purpose of the study is to evaluate the effect of kidney function on pharmacokinetics and pharmacodynamics of DWP16001 following single and multiple oral doses in type 2 diabetes patients with normal kidney function and renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 19 years at the time of screening test
* Body weight of ≥ 50.0 kg to ≤ 90.0 with a body mass index (BMI) of ≥ 20.0 to ≤ 45.0
* Have been diagnosed with type 2 diabetes

Exclusion Criteria:

* Have clinically uncontrolled or unstable hepatic, neurological, immune system, respiratory, hemato-oncology, cardiovascular, or psychiatric disorder (subject with chronic disease such as hypertension, diabetes, and hyperlipidemia that is well controlled or stable is eligible to participate in the study based on investigator's judgement)
* History of gastrointestinal diseases, dialysis, kidney transplantation, HIV, hepatitis B or C, acute or chronic infection, recent diabetic ketoacidosis, or gastrointestinal surgery that may affect the absorption of the study drug
* Received SGLT2 inhibitors or drugs of thiazolidinedione class within 6 weeks of scheduled IP administration day
* Clinical laboratory test values are outside the accepted normal range at screening

  * AST (SGOT), ALT (SGPT) > 2 x the upper limit of normal
  * Repeatedly confirmed QTc interval > 450 ms
* Sitting systolic blood pressure < 80 mmHg or > 180 mmHg or sitting diastolic blood pressure < 60 mmHg or > 110 mmHg after resting for more than 3 minutes
* Other exclusive inclusion criteria, as defined in the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | on Days 1 to 4 at selected time points
Concentration-time curve [AUC] | on Days 1 to 4 at selected time points
Urine glucose (g/day) | on Days -1 to 4
  Cummulative by time
Concentration of serum glucose | on Days 1 to 4 at selected time points

IPD SHARING:
Plan to Share IPD: No